CLINICAL TRIAL: NCT00021307
Title: Phase I/II Trial Of Temozolomide And Carboplatin In Recurrent Glioblastoma Multiforme
Brief Title: Temozolomide Plus Carboplatin in Treating Patients With Recurrent Glioblastoma Multiforme
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study not activated.
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: FCCC-01004; CDR0000068768 (Registry Identifier: PDQ (Physician Data Query)); NCI-G01-1981
Record Dates: First submitted 2001-07-11; First posted 2004-01-14 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carboplatin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: carboplatin
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of temozolomide plus carboplatin in treating patients who have recurrent glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose (MTD) of temozolomide and carboplatin in patients with recurrent glioblastoma multiforme. II. Determine the toxic effects of this regimen in these patients. III. Determine the pharmacokinetics of this regimen in these patients. IV. Determine the potential of either a pharmacokinetic or pharmacodynamic-mediated drug interaction in patients treated with this regimen. V. Determine the objective response rate and stabilization rate in patients treated with this regimen at the MTD. VI. Determine the acute and long-term toxic effects of this regimen at the MTD in these patients. VII. Determine the time to tumor progression and survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study. Patients are stratified according to age (under 50 vs 50 and over), ECOG performance status (0 vs 1-2), and prior therapy with carmustine or lomustine (yes vs no). Patients receive carboplatin IV over 30 minutes on day 1 and oral temozolomide on days 1-5. Treatment repeats every 4 weeks for a total of 6 courses in the absence of disease progression or unacceptable toxicity. Patients with stable or responsive disease may receive 6 additional courses of temozolomide. Cohorts of 1-6 patients receive escalating doses of carboplatin and temozolomide until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Additional patients are treated at the MTD.

PROJECTED ACCRUAL: Approximately 3-30 patients will be accrued for phase I of this study. A total of 16-58 patients will be accrued for phase II of this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed recurrent glioblastoma multiforme Measurable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: At least 12 weeks Hematopoietic: Granulocyte count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin at least 10.0 g/dL Hepatic: Bilirubin no greater than 1.5 times normal SGOT no greater than 3 times upper limit of normal Renal: Creatinine clearance greater than 50 mL/min Cardiovascular: No myocardial infarction within the past 6 months No congestive heart failure requiring therapy Other: HIV negative No active or uncontrolled infection No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix No frequent vomiting No medical condition that would interfere with oral medication intake (e.g., partial bowel obstruction) No known or suspected psychiatric disorder that would preclude study No other severe concurrent disease that would preclude study Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for at least 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent sargramostim (GM-CSF) No concurrent prophylactic filgrastim (G-CSF) Chemotherapy: No prior temozolomide No prior platinum-based chemotherapy Endocrine therapy: Not specified Radiotherapy: Not specified Surgery: Recovered from prior major surgery No more than 2 weeks since prior subtotal tumor resection Other: Recovered from prior therapy No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jon Glass, MD, Study Chair — Fox Chase Cancer Center